CLINICAL TRIAL: NCT04562545
Title: Effect of Incremental Versus Maximum Bite Advancement in Class II Subjects Using Twin Block Appliance : Randomized Clinical Trials
Brief Title: Twin Block Appliance in Incremental Versus Maximum Bite Advancement in Skeletal Class II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Khaled Mohamed Ali Hussein, Post Graduate Student, Department of Orthodontics, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD-CU-2020-09-08
Record Dates: First submitted 2020-09-08; First posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Mandibular Retrognathism; Mandibular Hypoplasia
Keywords: Twin Block; Bite Advancement; Growth Modification
MeSH Terms: conditions — Micrognathism

STUDY DESIGN:
Intervention Model Description: Type: Two arm, parallel, randomized clinical trial. allocation ratio 1:1 framework: superiority
Who Masked: Outcomes Assessor
Masking Description: Assessor will carry out measurements blindly on pre-operative and post-operative radio-graphs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maximum Bite Advancement (Active Comparator)
  Interventions: Device: Twin Block Appliance set to maximum bite
- Incremental Bite Advancement (Experimental)
  Interventions: Device: Modified Twin Block

INTERVENTIONS:
Device: Modified Twin Block — a modified twin block design including jack screws to facilitate incemental advancement
  Arms: Incremental Bite Advancement
Device: Twin Block Appliance set to maximum bite — a traditional twin block set to maximum bite advancement at start of treatment
  Arms: Maximum Bite Advancement

SUMMARY:
The aim of this study is to compare to different protocols to treat Class II malocclusion in growing subjects using the twin block appliance

DETAILED DESCRIPTION:
* Patients will be clinically and radio-graphically examined for eligibility
* Eligible patients will be randomly assigned to one of two groups:

  * Control Group: Twin Block Appliance fabricated to Maximum Bite Advancement group
  * Intervention Group: Twin Block Appliance fabricated for Incremental Bite Advancement group
* Records will be taken and impressions will be made and poured. In the control group, bite registration will be made with maximum mandibular advancement. In the intervention group, bite registration is made to habitual bite to make a modified twin block.
* Patients will be recalled every 6 weeks for 8 months for monitoring and reactivation of the appliance.

ELIGIBILITY:
Inclusion Criteria:

* Growing Female Patient
* Skeletal Class II Malocclusion due to deficient mandible
* Overjet of 7 to 10 mm
* Short or normal vertical facial pattern
* No previous orthodontic nor orthopedic treatment

Exclusion Criteria:

* Syndromes or Chronic Illness
* Skeletal Class II Malocclusion due to excessive maxilla
* Vertical skeletal growth pattern
* Habits

Ages: 9 Years to 13 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — biological growing female
Enrollment: 24 (Estimated)
Dates: Start 2020-09-15 (Estimated); Primary Completion 2021-09-15 (Estimated); Study Completion 2021-09-15 (Estimated)

PRIMARY OUTCOMES:
To asses Skeletal and dentoalveolar changes in Mandible | 8 Months
  Cone Beam CT will be taken before and after active treatment, 3D Cephalometric analysis will be conducted on the Cone Beam to asses Skeletal and Dentoalvoelar changes in mandible.
  - changes that will be assesed include ( mandibular base length / mandibular antero posterior position in relation to cranial base/ Condylar position / lower incisor inclination to mandibular plane)
To asses patient compliance | 8 months
  patient will answer a questionnaire at end of treatment

SECONDARY OUTCOMES:
To asses Skeletal and dentoalveolar changes in Maxilla | 8 months
  * Cone Beam CT will be taken before and after active treatment, 3D Cephalometric analysis will be conducted on the Cone Beam to asses Skeletal and Dentoalvoelar changes in maxilla
  * Changes that will be assesed include ( maxillary base length / maxillary base antero posterior position in relation to cranial base / incisor inclination to palatial plane)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
no plan to share data

REFERENCES:
- [Background] DeVincenzo JP, Winn MW. Orthopedic and orthodontic effects resulting from the use of a functional appliance with different amounts of protrusive activation. Am J Orthod Dentofacial Orthop. 1989 Sep;96(3):181-90. doi: 10.1016/0889-5406(89)90454-x. PMID 2773861
- [Background] Banks P, Wright J, O'Brien K. Incremental versus maximum bite advancement during twin-block therapy: a randomized controlled clinical trial. Am J Orthod Dentofacial Orthop. 2004 Nov;126(5):583-8. doi: 10.1016/j.ajodo.2004.03.024. PMID 15520691